CLINICAL TRIAL: NCT03025919
Title: Using 2h-glycosuria Combined With Fasting Plasma Glucose , Advanced Glycation End-product Alone or in Combination With Fasting Plasma Glucose in Diabetes Screening in Chinese Natural Population
Brief Title: Evaluation of Innovated Screening Tools for Type 2 Diabetes Among Chinese Population(SENSIBLE STUDY I)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Zilin Sun, director physician, Zhongda Hospital
Other Study IDs: 2016YFC1305700s
Record Dates: First submitted 2017-01-11; First posted 2017-01-20 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Type II Diabetes Mellitus
Keywords: Advanced glycation end-product; Glycosuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glycosuria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Evaluation of using 2h-UG combined with FPG, AGEsP alone or in combination with FPG in diabetes screening in Chinese natural population

DETAILED DESCRIPTION:
Using the WHO criteria as the golden standard，drawing the ROC curve of 2h-UG combined with FPG, AGEsP alone or in combination with FPG，calculating the area under the ROC curve.

ELIGIBILITY:
Inclusion Criteria:

* 20~70 year old urban and rural residents;
* Volunteer to participate in this study and sign informed consent.

Exclusion Criteria:

-

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Natural Chinese population
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12

PRIMARY OUTCOMES:
area under the ROC curve | 6 months
  area under the ROC curve of different method of using 2h-UG combined with FPG, AGEsP alone or in combination with FPG in diabetes screening in Chinese natural population

SECONDARY OUTCOMES:
sensitivity and specificity of screening | 6 months
  Using WHO criteria as golden standard,sensitivity and specificity of using 2h-UG combined with FPG, AGEsP alone or in combination with FPG in diabetes screening in Chinese natural population

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Zhongda Hospital, Institute of Diabetes, Southeast University, Nanjing, Jiangsu, China